CLINICAL TRIAL: NCT02252237
Title: Study of Pharmacokinetic Variability of Glucocorticoids in Children
Brief Title: Pharmacokinetics of Glucocorticoids in Children (GLUCOPED)
Acronym: GLUCOPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A00987-40
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Children Receiving Prednisone or Prednisolone or Methylprednisolone or Hydrocortisone
Keywords: Prednisone; Prednisolone; Methylprednisolone; Glucocorticoids; pharmacokinetics; hydrocortisone
MeSH Terms: interventions — Pharmacogenomic Variants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal cell collection swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with glucocorticoids: Children receiving Prednisone or Prednisolone or Methylprednisolone Pharmacokinetic
  Interventions: Biological: Pharmacokinetic

INTERVENTIONS:
Biological: Pharmacokinetic — Blood sample of 2 ml at enrolment and then at following visits. Buccal cell collection swab

SUMMARY:
The purpose of this study is to determine individual susceptibility factors (drug interactions, genetic factors such as enzyme polymorphism…) to explain wide interindividual variability towards corticosteroids (prednisone, prednisolone, methylprednisolone, hydrocortisone) in children, which could establish a base for therapeutic monitoring.

DETAILED DESCRIPTION:
Corticosteroids are widely used in children. A large interindividual variability exists concerning both efficacity and tolerance. Pharmacokinetic is poorly known.

A knowledge of individual susceptibility factors would allow to better adapt therapy in each case.

Drugs evaluated here are used in routine care in children and will be prescribed according to department practices concerning treated disease. Medical checks will be done during usual follow-up. Several features will be collected: reason of treatment, drug chosen and prescription modalities, observance, concomitant treatments, side effects, clinical examination, photography, score… Blood samples will be performed at different interval during usual biological follow-up. Three samples per patient will be required for pharmacokinetic and pharmacogenetic.

170 children under prednisone/prednisolone,130 under methylprednisolone, and 100 children under hydrocortisone will be recruited in four pediatric medical departments: immuno-hematology, nephrology,dermatology, and pediatric neurology.

ELIGIBILITY:
Inclusion Criteria:

* receiving Prednisone or Prednisolone or Methylprednisolone or hydrocortisone
* recruited in Immuno-hematological unit, dermatological unit, in pediatric nephrological unit, pediatric intensive care unit, or pediatric neurology unit
* parental agreement

Exclusion Criteria:

* parental refusal
* inability to take a blood sample
* inhaled corticoids intake in the 3 previous days
* topical corticoids intake in the 3 previous days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children receiving glucocorticoids (Prednisone or Prednisolone or Methylprednisolone or hydrocortisone) are recruited in Immuno-hematological unit, dermatological unit, in pediatric nephrological unit, pediatric intensive care unit, or pediatric neurology unit
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetic parameter for Prednisone, Prednisolone, Methylprednisolone, hydrocortisone | 24 months
  Assessed by:
  * Volume of distribution of creatinine
  * Creatinine clearance

SECONDARY OUTCOMES:
Side effects | 24 months
  Ferryman and Gallwey score
Side effects | 24 months
  Dermaphot® score
Analysis of genetic polymorphism of proteins taking part in glucocorticoids metabolism | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Tréluyer, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Necker, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jamroziak K, Mlynarski W, Balcerczak E, Mistygacz M, Trelinska J, Mirowski M, Bodalski J, Robak T. Functional C3435T polymorphism of MDR1 gene: an impact on genetic susceptibility and clinical outcome of childhood acute lymphoblastic leukemia. Eur J Haematol. 2004 May;72(5):314-21. doi: 10.1111/j.1600-0609.2004.00228.x. PMID 15059065
- [Background] Gatti G, Perucca E, Frigo GM, Notarangelo LD, Barberis L, Martini A. Pharmacokinetics of prednisone and its metabolite prednisolone in children with nephrotic syndrome during the active phase and in remission. Br J Clin Pharmacol. 1984 Apr;17(4):423-31. doi: 10.1111/j.1365-2125.1984.tb02367.x. PMID 6721988
- [Background] Miller PF, Bowmer CJ, Wheeldon J, Brocklebank JT. Pharmacokinetics of prednisolone in children with nephrosis. Arch Dis Child. 1990 Feb;65(2):196-200. doi: 10.1136/adc.65.2.196. PMID 2317067
- [Background] Petersen KB, Jusko WJ, Rasmussen M, Schmiegelow K. Population pharmacokinetics of prednisolone in children with acute lymphoblastic leukemia. Cancer Chemother Pharmacol. 2003 Jun;51(6):465-73. doi: 10.1007/s00280-003-0602-3. Epub 2003 Apr 16. PMID 12698270
- [Background] Faure C, Andre J, Pelatan C, Munck A, Giraud M, Cezard JP, Jacqz-Aigrain E. Pharmacokinetics of intravenous methylprednisolone and oral prednisone in paediatric patients with inflammatory bowel disease during the acute phase and in remission. Eur J Clin Pharmacol. 1998 Sep;54(7):555-60. doi: 10.1007/s002280050512. PMID 9832298
- [Result] de Truchis C, Bouazza N, Foissac F, Charbit M, Dehoux L, Lui G, Ribot M, Briand N, Zheng Y, Treluyer JM, Boyer O. Prednisolone pharmacokinetics after oral prednisone administration in paediatric patients with kidney transplant. Br J Clin Pharmacol. 2023 May;89(5):1532-1540. doi: 10.1111/bcp.15610. Epub 2022 Dec 12. PMID 36510685